CLINICAL TRIAL: NCT06910930
Title: Impact of Muscle Training Device on Non-Severe OSA: A Randomized Controlled Study
Brief Title: Impact of Muscle Training Device on Non-Severe OSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University Hospital (Other)
Responsible Party: Principal Investigator, Naphitchaya Wiriya, Naphitchaya Wiriya, MD., Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MTU-EC-IM-0-293/67
Record Dates: First submitted 2025-03-19; First posted 2025-04-04 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: OSA; Obstructive Sleep Apnea
Keywords: Device; EMST; Powerbreathe; didgeridoo; didgeriTU; Expiratory muscle exercise; reverse CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DidgeriTU (Active Comparator): patients with non severe OSA using DidgeriTU device
  Interventions: Device: DidgeriTU
- sham device (Sham Comparator): Patients with non severe OSA receive a device that look alike didgeriTU but without resistance plate
  Interventions: Device: Sham device

INTERVENTIONS:
Device: DidgeriTU — the study device that immitate the principle of didgeridoo for expiratory muscle exercise
  Arms: DidgeriTU
Device: Sham device — a device that look alike DidgeriTU but without resistance plate
  Arms: sham device

SUMMARY:
The goal of this clinical trial is to test for the efficacy of the newly invented device #DidgeriTU with non-severe obstructive sleep apnea. The main question it aims to answer is:

• Can DidgeriTU reduce apnea events in patients with non-severe obstructive sleep apnea? Researchers will compare DidgeriTU with a sham device to see how the apnea event has changed.

Participants will:

* Use DidgeriTU or sham device for 3 month
* Do an online questionnaire once a month during the study
* Home sleep test, lung function test, and tongue strength test at the start and end of the study

DETAILED DESCRIPTION:
Previously, in Switzerland, an aboriginal musical instrument, the Didgeridoo, was taught to patients with OSA. It has been proven to be effective in reducing apnea events.

Our newly invented instrument, DidgeriTU, adopts the Didgeridoo principle for expiratory muscle exercise to reduce apnea events.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with mild to moderate obstructive sleep apnea.
* Age 18 years or older.
* Patients voluntarily consent to provide information for research purposes.

Exclusion Criteria:

* Patients with an average apnea-hypopnea index (AHI) of <4 or >29 events per hour after repeated diagnosis using a home sleep apnea test.
* Patients who refused to cease using CPAP during the study process
* Patients with a history of chronic lung disease.
* Elderly patients with neurological conditions that impair cognitive function, such as dementia, stroke, or psychiatric disorders.
* Patients taking medications that may affect muscle function within 3 months before the start of the study.
* Patients with hypothyroidism or other conditions that may affect muscle function.
* Patients who consume alcohol at a moderate level or higher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Change of apnea event after DidgeriTU usage compared with sham device | 3 months
  Participants with a known history of non-severe obstructive sleep apnea will repeat the home sleep apnea test. The study will include patients with non-severe OSA(Apnea-hypopnea index 5-29/hr) from HSAT. After the usage of DidgeriTU or sham device for 3 months, the participant will repeat HSAT to explore the change of AHI after DidgeriTU use compared with sham device.

SECONDARY OUTCOMES:
Change of OSA severity after the usage of DidgeriTU comparing with sham device | 3 months
  Participants with a known history of non-severe obstructive sleep apnea will repeat the home sleep apnea test. The study will include patients with non-severe OSA(Apnea-hypopnea index 5-29/hr.) from HSAT and categorize patients with AHI 5-14/hr as mild OSA, AHI 15-29/hr as moderate OSA. After the usage of DidgeriTU or sham device for 3 months, the participant will repeat HSAT to explore the change of OSA severity after DidgeriTU use compared with sham device.
Change in Epworth sleepiness scale after the usage of DidgeriTU comparing with sham device | 3 months
  The participants' daytime sleepiness will be evaluated at the beginning of the study by the Thai version of the Epworth sleepiness scale then followed up with an online questionnaire every month until the end of the study. The total ESS score ranges from 0 to 24, with higher scores indicating greater daytime sleepiness. The change in ESS in patients using DidgeriTU will be compared with patients using sham devices.
Change of maximum inspiratory pressure; MIP after DidgeriTU usage comparing with sham device | 3 months
  The participants' maximum inspiratory pressure; MIP will be measured at the beginning and end of the study to compare the effect of DidgeriTU and sham device with inspiratory muscle which will be reported in cmH2O.
Change of maximum expiratory mouth pressure; MEP after DidgeriTU usage comparing with sham device | 3 months
  The participants' maximum expiratory mouth pressure; MEP will be measured at the beginning and end of the study to compare the effect of DidgeriTU and sham device with expiratory muscle which will be reported in cmH2O.
change in Pittsburg Sleep Quality Index; PSQI after DidgeriTU usage comparing with sham device | 3 months
  The participants' sleep quality will be evaluated at the beginning of the study by the Thai version of the Pittsburg sleep quality index then followed up with an online questionnaire every month until the end of the study. The global PSQI score ranges from 0 to 21, where lower scores indicate better sleep quality. The change in PSQI in patients using DidgeriTU will be compared with patients using sham devices.
Change of snoring frequency after DidgeriTU usage compared with a sham device | 3 months
  The snoring index (events/hour) will be recorded from HSAT at the beginning and end of the study. The change of snoring index from patients using DidgeriTU and sham device will be compared.
change of oxygenation during sleep after DidgeriTU usage comparing with sham device | 3 months
  The average oxygen saturation (%) will be recorded from HSAT at the beginning and end of the study. The change in average oxygen saturation from patients using DidgeriTU and sham device will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Thammasat University Hospital, Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: No